CLINICAL TRIAL: NCT06738927
Title: Otological Study of Facial Cleft Patients Over 10 Years of Age (Excluding Isolated Cleft Lip)
Brief Title: Otological Study of Facial Cleft Patients Over 10 Years of Age (Excluding Isolated Cleft Lip) (EFEOF)
Acronym: EFEOF
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC24.0229 - EFEOF
Record Dates: First submitted 2024-12-13; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-09

CONDITIONS: Serous Otitis; Tympanic Membrane Perforation; Retraction Pocket; Cholesteatoma; Otorrhea; Myringosclerosis; Tympanosclerosis; Audiometric Tests
Keywords: Serous otitis Tympanic membrane perforation Retraction pocket Cholesteatoma otorrhea Myringosclerosis Tympanosclerosis Audiometric tests; ENT; transtympanic ventilatory tubes.; cleft palate
MeSH Terms: conditions — Tympanic Membrane Perforation; Cholesteatoma; Myringosclerosis; Tympanosclerosis; Cleft Palate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Studies published on the placement of transtympanic ventilatory tubes in children with cleft palate show heterogeneous results, highlighting the need for a new study with strong statistical power and long-term follow-up to clarify the real benefits of this intervention.

Mirashrafi (2022) and Maina (2022), for example, emphasize the current uncertainties regarding the management of otitis media with effusion in children with cleft palate. Mirashrafi conducted a study on 40 children and found no significant difference between those with a complete cleft palate and those with an incomplete cleft palate in terms of middle ear status after the placement of transtympanic ventilatory tubes. Maina, in an ongoing review, identified a lack of consensus on the optimal management of chronic otitis media with effusion, with outcomes being varied and often of low methodological quality.

The absence of convincing evidence justifies the need for further research to establish clear guidelines. The objective is to study the otological status of patients based on the presence or absence of ENT surgical management involving the placement of transtympanic ventilatory tubes.

DETAILED DESCRIPTION:
The primary evaluation criterion will be ENT consultations:

Tympanic examination: Anatomical analysis of the tympanic membrane, assessing the presence or absence of:

Serous otitis Tympanic membrane perforation Retraction pocket Cholesteatoma Otorrhea Myringosclerosis Tympanosclerosis Audiometric tests: Assessment of auditory results from bone and air conduction curves for frequencies ranging from 250 to 4000 Hz, with analysis at every 250 Hz.

ELIGIBILITY:
Inclusion Criteria:

Presence of a facial cleft between 2004 and 2014 Minor and adult patients Followed up by ENT services at the University Hospital of Brest or Marseille

Exclusion Criteria:

Patients under legal protection (guardianship, curatorship, etc.) Refusal to participate Objection from one of the parents Isolated cleft lip No ENT follow-up

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals currently over 10 years old with an orofacial cleft (excluding isolated cleft lip).
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-12-12 (Estimated); Primary Completion 2024-12-12 (Estimated); Study Completion 2024-12-12 (Estimated)

PRIMARY OUTCOMES:
To study the otological status of patients based on the presence or absence of ENT surgical management involving the placement of transtympanic ventilatory tubes. | 01/01/2004 to 01/01/2014

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement